CLINICAL TRIAL: NCT00142987
Title: Efficacy of Tegaserod in Relieving the Symptoms of Female Patients With Irritable Bowel Syndrome (IBS), Excluding Those With Predominant Diarrhea IBS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHTF919A2417
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2008-01-28 (Estimated); Status verified 2008-01

CONDITIONS: IBS-C and IBS With Mixed Bowel Habits
Keywords: Tegaserod, IBS-C, women, mixed bowel habit
MeSH Terms: interventions — tegaserod

INTERVENTIONS:
Drug: Tegaserod

SUMMARY:
Recent literature has demonstrated that the group of IBS sufferers who experience mixed bowel habits may be more similar to IBS-C patients than IBS-D patients. This study will evaluate the efficacy and safety of tegaserod 6 mg b.i.d. in women with IBS and mixed bowel habits, excluding those with predominant diarrhea.

ELIGIBILITY:
Inclusion Criteria:

* women, outpatients, 18-65 years of age with IBS-C or IBS with mixed bowel habits
* In the 12 months preceding study entry, they had to have at least 12 weeks (not necessarily consecutive) of abdominal discomfort/pain with 2 out of 3 features: 1) relieved with defecation; 2) onset associated with a change in stool frequency; 3) onset associated with a change in form (appearance) of stool.
* Had to fulfill the following criteria (IBS questionnaire) during the last 3 months prior to study entry: abdominal discomfort or pain present during at least 3 weeks in the last 3 months, and at least two of the following: abdominal discomfort or pain gets better or stops after a bowel movement; change in bowel movement frequency when the abdominal discomfort or pain starts; change in bowel movement consistency when the abdominal discomfort or pain starts

Exclusion Criteria:

* IBS-D
* not reporting any constipation and diarrhea criteria
* evidence of structural abnormality of the gastrointestinal tract or diseases/conditions that affect bowel transit
* history of bowel obstruction, symptomatic gallbladder disease, suspected sphincter of Oddi dysfunction, or abdominal adhesions
* evidence of cathartic colon or history of laxative abuse

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult
Enrollment: 664
Dates: Start 2004-04; Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Weekly assessment of patient's overall satisfaction relief over 4 weeks of treatment of IBS symptoms

SECONDARY OUTCOMES:
Weekly assessment of patient's overall satisfaction relief.
Over 4 weeks of treatment and during each week improvment of abdominal discomfort pain, bloating, stool frequency, stool consitency, straining urgency.
During 4 week treatment period efficacy assessment in IBS-C subgroup and mixed IBS.
Assessment of safety and tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — East Hanover NJ